CLINICAL TRIAL: NCT01383226
Title: CT Enlarged Mediastinal/Hilar Lymph Nodes Not Visible on Chest X-ray in the Non Cancer Patient : Diagnosis and Clinical Implications Using Endobronchial or Esophageal Ultrasound Controlled Needle Aspiration E(B)US-NA
Brief Title: Linear Endosonography for the Assessment of Sarcoidosis Stage O
Acronym: LASSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S53313
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Lymphadenitis
Keywords: endosonography; enlarged thoracic lymph adenopathies; non-cancer patient
MeSH Terms: conditions — Lymphadenitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thoracic endosonography (Other): Thoracic endosonography, either endobronchial or esophageal ultrasound controlled needle aspiration, is a minimally invasive diagnostic technique.
  Interventions: Procedure: Thoracic endosonography

INTERVENTIONS:
Procedure: Thoracic endosonography — Thoracic endosonography is a minimal invasive diagnostic intervention

SUMMARY:
Patients are often referred for E(B)US examination and sampling of enlarged mediastinal and/or hilar lymph nodes that are not visible on a standard chest X-ray but are discovered by accident on CT scan performed outside the context of lung cancer or extrathoracic malignancies. Since CT scan is largely used and E(B)US is a minimally invasive technique, these cases are explored more frequently but so far nothing is known, however, on the prevalence of abnormal findings in EBUS sampling in this particular population and on the clinical implications (mainly therapeutical implications) of E(B)US findings.

DETAILED DESCRIPTION:
The primary aim is to assess the nature and prevalence of abnormal findings in samplings obtained during E(B)US-NA in the non-cancer patient with CT enlarged mediastinal/hilar lymph nodes that are not visible on chest X-ray. As secondary aims, the clinical implications of E(B)US-NA findings will be assessed, in particular the number of cases where a specific treatment is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to bronchoscopy for tissue diagnosis of discrete enlarged (≥10mm short axis diameter) mediastinal/hilar lymph nodes on CT scan that can be sampled by E(B)US-NA.

Exclusion Criteria:

* Abnormal chest X-ray showing hilar/mediastinal lymph nodes
* Patients with suspected lung cancer
* Patients with previous malignancy diagnosed and definitely treated less than 5 years previously or, if treated more than five years before but with subsequent evidence of recurrence less than 5 years previously.
* Patient with concomitant (suspected or confirmed) bronchopulmonary infection or treated with antibiotics within the 4 previous weeks
* Patients with a contraindication for bronchoscopy and tissue sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity | One year
  The primary aim is to assess the nature and prevalence of abnormal findings in samplings obtained during E(B)US-NA in the non-cancer patient with CT enlarged mediastinal/hilar lymph nodes that are not visible on chest X-ray.

SECONDARY OUTCOMES:
Clinical impact. | One year
  As secondary aims, the clinical implications of E(B)US-NA findings will be assessed, in particular the number of cases where a specific treatment is initiated.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe A Dooms, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Vincent Ninane, MD, PhD, Principal Investigator — Hopital Saint-Pierre Brussels
Locations (9):
- Belgium (9):
  - Middelheim Ziekenhuis, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - Hopital Saint-Pierre Bruxelles, Brussels
  - Centre Hospitalier Universitaire Charleroi, Charleroi
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven
  - Heilig Hart Ziekenhuis Roeselare, Roeselare
  - Sint-Elisabeth Ziekenhuis, Turnhout
  - Université Catholic Louvain, Woluwe